CLINICAL TRIAL: NCT04087759
Title: Phase 1, Open-label, Randomized Crossover Study in Healthy Adult Subjects to Assess the Relative Oral Bioavailability and Food Effect of Bedaquiline 100-mg Tablets Administered as Different Test Formulations Compared to the Commercial Tablet Formulation (F001)
Brief Title: A Study of Bedaquiline 100 Milligram (mg) Tablets Administered as Different Test Formulations Compared to the Commercial Tablet Formulation (F001) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108659; 2018-004306-26 (EudraCT Number); TMC207TBC1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence BAE (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral test tablet 1 under fasted condition (Treatment B) in period 1, followed by bedaquiline oral reference tablet under fasted condition (Treatment A) in period 2, thereafter will receive bedaquiline oral test tablet 1 under fed condition (Treatment E) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)
- Treatment Sequence CAF (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral test tablet 2 under fasted condition (Treatment C) in period 1, followed by bedaquiline oral reference tablet under fasted condition (Treatment A) in period 2, thereafter will receive bedaquiline oral test tablet II under fed condition (Treatment F) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)
- Treatment Sequence DAG (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral test tablet 3 under fasted condition (Treatment D) in period 1, followed by bedaquiline oral reference tablet under fasted condition (Treatment A) in period 2, thereafter will receive bedaquiline oral test tablet 3 under fed condition (Treatment G) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)
- Treatment Sequence ABE (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral reference tablet under fasted condition (Treatment A) in period 1, followed by bedaquiline oral test tablet 1 under fasted condition (Treatment B) in period 2, thereafter will receive bedaquiline oral test tablet 1 under fed condition (Treatment E) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)
- Treatment Sequence ACF (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral reference tablet under fasted condition (Treatment A) in period 1, followed by bedaquiline oral test tablet 2 under fasted condition (Treatment C) in period 2, thereafter will receive bedaquiline oral test tablet 2 under fed condition (Treatment F) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)
- Treatment Sequence ADG (Experimental): Participants will receive a single dose of bedaquiline in 3 subsequent sessions as bedaquiline oral reference tablet under fasted condition (Treatment A) in period 1, followed by bedaquiline oral test tablet 3 under fasted condition (Treatment D) in period 2, thereafter will receive bedaquiline oral test tablet 3 under fed condition (Treatment G) in period 3. Each treatment period will be separated with a washout period of at least 28 days.
  Interventions: Drug: Bedaquiline (Test formulation); Drug: Bedaquiline (Reference formulation)

INTERVENTIONS:
Drug: Bedaquiline (Test formulation) — Participants will receive bedaquiline orally.
  Other Names: JNJ-16175328
Drug: Bedaquiline (Reference formulation) — Participants will receive bedaquiline orally.
  Other Names: SIRTURO, TMC207

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of bedaquiline following administration of a single oral dose of 100 milligram (mg) equivalent (1*100 mg) given as different test tablet formulations compared to the administration of a single oral dose of 100 mg equivalent (1*100 mg) formulated as SIRTURO commercial tablet (formulation F001), under fasted conditions in healthy adult participants. Also, to assess the effect of a standardized breakfast on the rate and extent of absorption of bedaquiline compared to fasted conditions following administration of a single oral dose of 100 mg equivalent (1*100 mg) for each of the different test tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* A female participant must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 in each treatment period
* Contraceptive use by women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* Participant must have a blood pressure (BP); supine after at least 5 minutes rest) between 90 and 140 millimeter of mercury (mmHg) systolic, extremes included, and no higher than 90 mmHg diastolic at screening
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) performed at screening (results must be available on Day -1). If there are abnormalities participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must have a body mass index (BMI); weight per height square between 18.0 and 30.0 kilogram per meter square (kg/m^2) (extremes included) at screening. The minimum body weight must be 50.0 kg at screening

Exclusion Criteria:

* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has known allergies, hypersensitivity, or intolerance to bedaquiline or its excipients
* Participant has received an investigational drug or used an invasive investigational medical device within 30 days or within a period less than 10 times the drug's elimination half-life (whichever is longer), or participant has received a biological product within 3 months or within a period less than 5 elimination half-lives (whichever is longer) before the planned first intake of study drug
* Participant has a history of human immunodeficiency virus (HIV)-1 or HIV-2 infection, or tests positive for HIV-1 or -2 at screening
* Participant has previously been dosed with bedaquiline, either in single or multiple dose studies, or participant with a previous history of pulmonal infection with Mycobacterium species

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Bedaquiline | Predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, and 672 hours postdose
  Cmax is the maximum observed analyte concentration.
Area Under the Analyte Concentration-time Curve from Time 0 to 72 Hours (AUC [0-72 hours]) of Bedaquiline | Predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, and 72 hours postdose
  AUC (0-72 hours) is area under the analyte concentration-time curve from time 0 to 72 hours, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC [0-last]) of Bedaquiline | Predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, and 672 hours postdose
  AUC (0-last) is area under the analyte concentration-time curve from time zero to the time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of Bedaquiline | Predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, 216, 264, 336, 504, and 672 hours postdose
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinity time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable concentration, and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 112 Days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment. Therefore, it can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency